CLINICAL TRIAL: NCT04615832
Title: F&P Toffee Full Face Mask Clinical Trial, NZ, 2020
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-284
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Positive Airway Pressure Therapy; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toffee Full Face Mask (Experimental): Toffee Full Face Mask: Full face mask for PAP therapy applied in a home environment for 2 weeks.
  Interventions: Device: Toffee Full Face Mask

INTERVENTIONS:
Device: Toffee Full Face Mask — Full face mask for PAP therapy applied in a home environment

SUMMARY:
This will be a prospective, multi-arm, randomized, and non-blinded clinical trial designed to evaluate the performance, comfort, and usability of the Toffee full face mask amongst participants who have been prescribed PAP therapy by a physician. This clinical trial will take place across three investigation sites with a sample of 45 participants.

DETAILED DESCRIPTION:
The purpose of this clinical investigation was to evaluate the performance, comfort and ease of use of the F&P Toffee Full Face Mask. The clinical investigation took place across three sites in order to recruit the required number of participants. The clinical investigation tested the mask on 44 participants, who were currently using a full face mask for PAP therapy.

This was a non-randomized non-blinded single intervention study. Informed consent was gathered from the 44 participants before demographic and baseline measurements were recorded. Participants were issued an appropriate fitting Toffee Full face mask for the two week at home trial.

After two weeks the participants returned the masks. At this visit device data was downloaded and participant questionnaires were completed.

ELIGIBILITY:
Inclusion Criteria:

* Persons who are ≥ 22 years of age
* Persons who weigh ≥ 66 lbs (30 kgs)
* Persons who have been prescribed PAP (APAP, BPAP or CPAP) therapy by a physician
* Persons who are compliant with PAP therapy for ≥ 4 hours per night for 70% of nights for at least two weeks prior to enrolment in the trial
* Persons who are currently using a full face mask
* Persons who have an IPAP pressure of < 30 cmH2O
* Persons who currently use a PAP therapy device with data recording capabilities
* Persons who are fluent in spoken and written English
* Persons who possess the capacity to provide informed consent

Exclusion Criteria:

* Persons who are intolerant to PAP therapy
* Persons who are required to use PAP therapy for more than 12 hours per day or for extensive periods other than sleep or naps
* Persons using nasal or nasal pillows masks
* Persons who possess, or suffer from, anatomical or physiological conditions which make PAP therapy inappropriate
* Persons who are pregnant or think they may be pregnant
* Persons who use a PAP therapy machine for the delivery of medicines, except supplemental O2
* Persons who currently have cold or flu like symptoms at the time of recruitment
* Persons who have tested positive for COVID-19 within the previous 28 days prior to enrolment

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavi Ogra, Principal Investigator — Fisher & Paykel Healthcare
Locations (3):
- New Zealand (3):
  - Hastings Memorial Hospital, Hastings, Hawkes Bay
  - Fisher & Paykel Healthcare, Auckland
  - Bowen Hospital, Wellington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Toffee Full Face Mask
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Toffee Full Face Mask
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 44

OUTCOME MEASURES:

1. Primary Outcome: Comfort - Subjective
Description: To assess the comfort of the mask as experienced by the participant. Comfort will be measured on a 4 point likert type scale (options: Very Uncomfortable, Uncomfortable, Comfortable, and Very Comfortable). Very Comfortable will be scored the highest and Very Uncomfortable will be scored the lowest. Different aspects of the mask such as cushion comfort, headgear comfort and overall comfort will be assessed using the same scale. Questions will be asked on a questionnaire and further qualitative responses will be captured during an interview.
Time Frame: Assessed 2 weeks after mask fitting
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Full Face Mask
Number analyzed (Participants) | 44
Participants
  Very comfortable | 18
  Comfortable | 23
  Uncomfortable | 2
  Very uncomfortable | 1

2. Primary Outcome: Usability
Description: To assess the ease of use of the mask as experienced by the participant. Questions regarding the freedom of movement in bed will be asked using a 4 point likert type scale (options: Very Difficult, Difficult, Easy, and Very Easy). Very Easy will be scored the highest and Very Difficult will be scored the lowest. Questions will be asked via a questionnaire with additional qualitative responses captured during an interview.
Time Frame: Assessed 2 weeks after mask fitting
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Full Face Mask
Number analyzed (Participants) | 44
Participants
  Very easy | 19
  Easy | 23
  Difficult | 2
  Very difficult | 0

3. Primary Outcome: Seal Performance
Description: To assess the sealing performance of the mask when used in a home environment. Questions regarding the seal performance will be asked using a 4 point likert type scale (options: Very poor, Poor, Good, and Very good). Very good will be scored the highest and Very poor will be scored the lowest.
Time Frame: Assessed 2 weeks after mask fitting
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Full Face Mask
Number analyzed (Participants) | 44
Participants
  Very good | 25
  Good | 15
  Poor | 4
  Very poor | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the 2 week duration of the study period.
Arm/Group | Toffee Full Face Mask
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 10/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toffee Full Face Mask (N=44)
Nasal soreness (Injury, poisoning and procedural complications) | 1 (1) — Due to previous nasal surgery. Not related, resolved no sequel.
Broken ankle (Injury, poisoning and procedural complications) | 1 (1) — Unrelated, resolved no sequel
Nasal compression (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Related, ongoing at study end.
Knee pain (Injury, poisoning and procedural complications) | 1 (1) — From previous surgery. Not related, resolved with sequel.
Left shoulder pain (Injury, poisoning and procedural complications) | 1 (1) — After strain. Not related, ongoing at study end.
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly related, resolved no sequel
Eye irritation (Eye disorders) | 2 (2) — Following up.
Mouth abscess (Psychiatric disorders) | 1 (1) — Stress induced. Not related, resolved no sequel.
Mouth Ulcer (Gastrointestinal disorders) | 1 (1) — Not related, ongoing at study end.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04615832/Prot_SAP_000.pdf